CLINICAL TRIAL: NCT06253559
Title: Clinical and Pathological Characteristics of Women With Ovarian Cancers, A National, Retrospective Cross-Sectional Study in Syria During the War
Brief Title: Clinical and Pathological Characteristics of Women With Ovarian Cancers in Syria
Status: Completed | Type: Observational
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Other Study IDs: TishreenU -Ovarian Cancer
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ovarian cancer patients: all ovarian cancer patients that meet the criteria of the study

SUMMARY:
the goal of this observational study is to describe ovarian cancer epidemiology and characteristics in Syrian women, especially during the war to do more research in the future about the risk factors of ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer (OC) is the eighth most common cause of death worldwide, and current studies show that the death numbers caused by it will rise dramatically in the coming years. As the epidemiological features of the cancer may vary, studying these different characteristics can help us improve treatment outcomes and add preventive measures. In addition, giving special attention to these features in developing countries, or countries undergoing crisis, will help us understand the associated risk factors in these regions.

ELIGIBILITY:
Inclusion Criteria:

* female adult (age ≥18 years)
* primary ovarian malignancy

Exclusion Criteria:

* less than 18 years old
* women who have benign tumors or metastatic ovarian cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all women with ovarian cancer, with age ≥18 years,who have primary ovarian malignancy and underwent surgical or non-surgical treatment.
  the data recorded from records of the Departments of Gynecology and Oncology at Tishreen University Hospital in Latakia, Al-Bairouni University Hospital in Damascus, and Ibn Rushd Hospital in Aleppo, which are the 3 major hospitals in Syria that admit and treat patients with ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
age | jan 2017 - july 2021
  the age of patients at the time of diagnosis
ovarian cancer grade | jan 2017 - july 2021
  ovarian cancer grades frequency among patients
histological type of ovarian cancer | jan 2017 - july 2021
  detect the most common type of ovarian cancer
sideness of ovarian cancer | jan 2017 - july 2021
  study the frequency of bilateral or unilateral ovarian cancer
Cancer Antigen-125 | jan 2017 - july 2021
  Cancer Antigen-125 levels, if they are normal or high in ovarian cancer.
Treatment | jan 2017 - july 2021
  detect if the patient underwent surgery or chemotherapy or the both
symptoms of ovarian cancer | jan 2017 - july 2021
  detect symptoms of disease at diagnosis time

CONTACTS AND LOCATIONS:
Overall Officials: Apelian, Principal Investigator — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided
data can be shared upon your request

REFERENCES:
- [Background] Zheng G, Yu H, Kanerva A, Forsti A, Sundquist K, Hemminki K. Familial risks of ovarian cancer by age at diagnosis, proband type and histology. PLoS One. 2018 Oct 3;13(10):e0205000. doi: 10.1371/journal.pone.0205000. eCollection 2018. PMID 30281663
- [Background] Wentzensen N, Poole EM, Trabert B, White E, Arslan AA, Patel AV, Setiawan VW, Visvanathan K, Weiderpass E, Adami HO, Black A, Bernstein L, Brinton LA, Buring J, Butler LM, Chamosa S, Clendenen TV, Dossus L, Fortner R, Gapstur SM, Gaudet MM, Gram IT, Hartge P, Hoffman-Bolton J, Idahl A, Jones M, Kaaks R, Kirsh V, Koh WP, Lacey JV Jr, Lee IM, Lundin E, Merritt MA, Onland-Moret NC, Peters U, Poynter JN, Rinaldi S, Robien K, Rohan T, Sandler DP, Schairer C, Schouten LJ, Sjoholm LK, Sieri S, Swerdlow A, Tjonneland A, Travis R, Trichopoulou A, van den Brandt PA, Wilkens L, Wolk A, Yang HP, Zeleniuch-Jacquotte A, Tworoger SS. Ovarian Cancer Risk Factors by Histologic Subtype: An Analysis From the Ovarian Cancer Cohort Consortium. J Clin Oncol. 2016 Aug 20;34(24):2888-98. doi: 10.1200/JCO.2016.66.8178. Epub 2016 Jun 20. PMID 27325851
- [Background] Yuan R, Zhang C, Li Q, Ji M, He N. The impact of marital status on stage at diagnosis and survival of female patients with breast and gynecologic cancers: A meta-analysis. Gynecol Oncol. 2021 Sep;162(3):778-787. doi: 10.1016/j.ygyno.2021.06.008. Epub 2021 Jun 16. PMID 34140180
- [Background] Torre LA, Trabert B, DeSantis CE, Miller KD, Samimi G, Runowicz CD, Gaudet MM, Jemal A, Siegel RL. Ovarian cancer statistics, 2018. CA Cancer J Clin. 2018 Jul;68(4):284-296. doi: 10.3322/caac.21456. Epub 2018 May 29. PMID 29809280
- [Background] Shanmughapriya, S., Senthilkumar, G., Arun, S., Das, B. C., & Natarajaseenivasan, K. (2016). Risk factors for epithelial ovarian carcinoma in India: A case control study in low-incidence population. International Journal of Cancer Research, 12(1), 61-68. https://doi.org/10.3923/IJCR.2016.61.68
- [Background] Reid BM, Permuth JB, Sellers TA. Epidemiology of ovarian cancer: a review. Cancer Biol Med. 2017 Feb;14(1):9-32. doi: 10.20892/j.issn.2095-3941.2016.0084. PMID 28443200
- [Background] Prat J. Ovarian carcinomas: five distinct diseases with different origins, genetic alterations, and clinicopathological features. Virchows Arch. 2012 Mar;460(3):237-49. doi: 10.1007/s00428-012-1203-5. Epub 2012 Feb 10. PMID 22322322
- [Background] Parazzini F, Franceschi S, La Vecchia C, Fasoli M. The epidemiology of ovarian cancer. Gynecol Oncol. 1991 Oct;43(1):9-23. doi: 10.1016/0090-8258(91)90003-n. PMID 1959794
- [Background] Momenimovahed Z, Tiznobaik A, Taheri S, Salehiniya H. Ovarian cancer in the world: epidemiology and risk factors. Int J Womens Health. 2019 Apr 30;11:287-299. doi: 10.2147/IJWH.S197604. eCollection 2019. PMID 31118829
- [Background] Meena RK, Syed NA, Sheikh ZA, Guru FR, Mir MH, Banday SZ, Mp AK, Parveen S, Dar NA, Bhat GM. Patterns of Treatment and Outcomes in Epithelial Ovarian Cancer: A Retrospective North Indian Single-Institution Experience. JCO Glob Oncol. 2022 Nov;8:e2200032. doi: 10.1200/GO.22.00032. PMID 36332174
- [Background] McCluggage WG. Morphological subtypes of ovarian carcinoma: a review with emphasis on new developments and pathogenesis. Pathology. 2011 Aug;43(5):420-32. doi: 10.1097/PAT.0b013e328348a6e7. PMID 21716157
- [Background] Lukanova A, Kaaks R. Endogenous hormones and ovarian cancer: epidemiology and current hypotheses. Cancer Epidemiol Biomarkers Prev. 2005 Jan;14(1):98-107. PMID 15668482
- [Background] the World Cancer Research Fund (WCRF), worldwide cancer data., 2020; https://www.wcrf.org/cancer-trends/worldwide-cancer-data/ )
- [Background] Lima MA, Dos Santos L, Turri JA, Nonogaki S, Buim M, Lima JF, de Jesus Viana Pinheiro J, Bueno de Toledo Osorio CA, Soares FA, Freitas VM. Prognostic Value of ADAMTS Proteases and Their Substrates in Epithelial Ovarian Cancer. Pathobiology. 2016;83(6):316-26. doi: 10.1159/000446244. Epub 2016 Jul 1. PMID 27359117
- [Background] Hayat MJ, Howlader N, Reichman ME, Edwards BK. Cancer statistics, trends, and multiple primary cancer analyses from the Surveillance, Epidemiology, and End Results (SEER) Program. Oncologist. 2007 Jan;12(1):20-37. doi: 10.1634/theoncologist.12-1-20. PMID 17227898
- [Background] Funston G, Hamilton W, Abel G, Crosbie EJ, Rous B, Walter FM. The diagnostic performance of CA125 for the detection of ovarian and non-ovarian cancer in primary care: A population-based cohort study. PLoS Med. 2020 Oct 28;17(10):e1003295. doi: 10.1371/journal.pmed.1003295. eCollection 2020 Oct. PMID 33112854
- [Background] Chornokur G, Amankwah EK, Schildkraut JM, Phelan CM. Global ovarian cancer health disparities. Gynecol Oncol. 2013 Apr;129(1):258-64. doi: 10.1016/j.ygyno.2012.12.016. Epub 2012 Dec 22. PMID 23266352
- [Background] Arora T, Mullangi S, Vadakekut ES, Lekkala MR. Epithelial Ovarian Cancer. 2024 May 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK567760/ PMID 33620837
- [Background] Arora N, Talhouk A, McAlpine JN, Law MR, Hanley GE. Long-term mortality among women with epithelial ovarian cancer: a population-based study in British Columbia, Canada. BMC Cancer. 2018 Oct 25;18(1):1039. doi: 10.1186/s12885-018-4970-9. PMID 30359249
- [Background] Andrews L, Mutch DG. Hereditary Ovarian Cancer and Risk Reduction. Best Pract Res Clin Obstet Gynaecol. 2017 May;41:31-48. doi: 10.1016/j.bpobgyn.2016.10.017. Epub 2017 Jan 17. PMID 28254144
- [Background] Zhang S, Cheng C, Lin Z, Xiao L, Su X, Zheng L, Mu Y, Liao M, Ouyang R, Li W, Ma J, Cai J, Liu L, Wang D, Zeng F, Liu J. The global burden and associated factors of ovarian cancer in 1990-2019: findings from the Global Burden of Disease Study 2019. BMC Public Health. 2022 Jul 30;22(1):1455. doi: 10.1186/s12889-022-13861-y. PMID 35907822
- [Background] Saki S, Ali NR, Saki SS, AlRabeea ZS, AlRemeithi FN, Carrick FR, Abdulrahman M. Barriers to healthcare seeking, beliefs about ovarian cancer and the role of socio-economic position. A cross-sectional multilevel study in Dubai, a multicultural society. J Public Health Res. 2021 Mar 24;10(3):2073. doi: 10.4081/jphr.2021.2073. PMID 33759446
- [Background] Ovarian cancer statistics | World Cancer Research Fund International. (n.d.). Retrieved May 19, 2023, from https://www.wcrf.org/cancer-trends/ovarian-cancer-statistics/
- [Background] Syria crisis . (n.d.). Retrieved May 19, 2023, from https://www.who.int/emergencies/situations/syria-crisis
- [Background] Holschneider CH, Berek JS. Ovarian cancer: epidemiology, biology, and prognostic factors. Semin Surg Oncol. 2000 Jul-Aug;19(1):3-10. doi: 10.1002/1098-2388(200007/08)19:13.0.co;2-s. PMID 10883018
- [Background] Gaona-Luviano P, Medina-Gaona LA, Magana-Perez K. Epidemiology of ovarian cancer. Chin Clin Oncol. 2020 Aug;9(4):47. doi: 10.21037/cco-20-34. Epub 2020 Jun 30. PMID 32648448
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Boussios S, Karathanasi A, Zakynthinakis-Kyriakou N, Tsiouris AK, Chatziantoniou AA, Kanellos FS, Tatsi K. Ovarian carcinosarcoma: Current developments and future perspectives. Crit Rev Oncol Hematol. 2019 Feb;134:46-55. doi: 10.1016/j.critrevonc.2018.12.006. Epub 2018 Dec 24. PMID 30771873
- [Background] Atallah GA, Abd Aziz NH, Teik CK, Shafiee MN, Kampan NC. New Predictive Biomarkers for Ovarian Cancer. Diagnostics (Basel). 2021 Mar 7;11(3):465. doi: 10.3390/diagnostics11030465. PMID 33800113
- [Background] Yoneda A, Lendorf ME, Couchman JR, Multhaupt HA. Breast and ovarian cancers: a survey and possible roles for the cell surface heparan sulfate proteoglycans. J Histochem Cytochem. 2012 Jan;60(1):9-21. doi: 10.1369/0022155411428469. PMID 22205677